CLINICAL TRIAL: NCT01027910
Title: Phase I/II Study of PCI-24781 in Combination With Doxorubicin for Treatment of Advanced Sarcomas Following Failure or Prior Anthracycline Therapy
Brief Title: PCI-24781 in Combination With Doxorubicin to Treat Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Pharmacyclics LLC. (Industry)
Responsible Party: Principal Investigator, Edwin Choy, MD, Principle Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-352
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Sarcoma
Keywords: PCI-24781; doxorubicin
MeSH Terms: conditions — Sarcoma | interventions — abexinostat; Doxorubicin; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCI-24781 without mandated GCSF (Experimental): PCI-24781 in combination with doxorubicin without mandated GCSF
  Interventions: Drug: PCI-24781; Drug: Doxorubicin; Drug: GCSF
- PCI-24781 with mandated GCSF (Experimental): PCI-24781 in combination with doxorubicin with mandated GCSF
  Interventions: Drug: PCI-24781; Drug: Doxorubicin; Drug: GCSF

INTERVENTIONS:
Drug: PCI-24781 — Capsules taken orally for 5 consecutive days starting on Day 1 of each 3 week cycle
  Other Names: PCI24781
Drug: Doxorubicin — Administered intravenously on Day 4 of each 3 week cycle
  Other Names: Adriamycin
Drug: GCSF — Administered on Day 5 of each 3 weeks cycle in Arm 1 if determined to be clinically indicated, and in all patients enrolled into Arm 2
  Other Names: Neupogen

SUMMARY:
The purpose of this research study is to determine the safety and maximum tolerated dose of PCI-24781 that can be given safely with doxorubicin (phase I) and the safety and efficacy of PCI-24781 when used in combination with doxorubicin (phase II) in patients with advanced sarcomas. The study drug, PCI-24781, is believed to regulate genes involved in tumor cell growth. The other study drug, doxorubicin, is considered a standard chemotherapeutic treatment for advanced sarcoma patients. We hypothesize that combining PCI-24781 with doxorubicin can overcome chemoresistance to doxorubicin.

DETAILED DESCRIPTION:
* In the phase I portion of the study, since we are looking for the highest dose of PCI-24781 that can be administered safely without severe or unmanageable side effects in participants that have advanced sarcoma, not everyone who participates in this research study will receive the same dose of PCI-24871.
* Each treatment cycle is 3 weeks (21 days). Participants will take capsules of PCI-24871 for five consecutive days starting on Day 1 of each 3 week cycle. On Day 4 of each cycle, participants will come to the clinic to receive doxorubicin intravenously.
* At specific time intervals, participants will return to the clinic for the following tests and procedures: physical examination, vital signs, blood tests, urine test, EKG, assessment of the tumor by CT scan, and an ECHO or MUGA.
* Participants may remain on the study for a maximum of 6 cycles (about 4-5 months). After the last cycle, as long as the participant is showing benefit, they may elect to continue taking PCI-24781 alone, in which case they will continue in this research study until there is evidence of their tumor growing.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed metastatic or unresectable sarcoma
* All participants must have received no more than a lifetime cumulative maximum dose of 300 mg/m2 or less of prior doxorubicin and no other anthracycline therapy.
* Participants must have measurable disease, defined as at least one unirradiated lesion that can be accurately measured in at least one dimension as 20mm or greater with conventional techniques or as 10mm or greater with spiral CT scan.
* ECOG performance status of 2 or less
* Ability to swallow oral capsules without difficulty
* Participants must have normal organ and marrow function as outlined in the protocol.
* Women of childbearing potential must have a negative serum/urine pregnancy test within 7 days prior to receiving the first dose of PCI-24781.
* An ECHO or MUGA demonstrating EF > 50% is required within 4 weeks prior to study drug administration.
* 18 years of age or older

Exclusion Criteria:

* Participants who have had immunotherapy, chemotherapy, experimental therapy or radiotherapy within 4 weeks before first day of study drug dosing or those who have not recovered to grade 1 or baseline from adverse events due to agents administered more than 4 weeks earlier.
* Participants who have previously received > 300 mg/m2 cumulative lifetime dose of doxorubicin, or who have received any other anthracycline chemotherapy.
* Major surgery within 4 weeks before first day of study drug dosing
* Participants with known central nervous system/brain metastases
* Participants receiving chronic corticosteroids > 20 mg prednisone equivalent per day for > 7 consecutive days (Topical, inhaled or nasal corticosteroids are permitted).
* Participants with any documented malabsorption syndromes or other conditions that may impair the absorption of PCI-24781 capsules.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants requiring concurrent therapeutic anticoagulation or have received therapeutic anticoagulation within 2 weeks of the first day of dosing.
* Risk factors for Torsades de Pointes, or use, within 4 weeks of starting study drug administration, of medications known to prolong QTc interval or that may be associated with Torsades de Pointes.
* QTc prolongation or other significant ECG abnormalities defined as 2nd degree AV block type II, 3rd degree AV block, or bradycardia.
* History of myocardial infarction, acute coronary syndromes, coronary angioplasty and/or coronary artery stenting within the past 6 months.
* For patients with history of major coronary artery disease in the judgement of the responsible physician, a cardiac stress test that demonstrates clinically significant abnormalities when performed within 28 days of first dose of study drug
* Pregnant or breastfeeding women
* Women of childbearing potential, or sexually active men unwilling to use adequate contraceptive protection during the course of the study
* HIV-positive individuals
* Other medical or psychiatric illness or organ dysfunction that, in the opinion of the investigator, would either compromise the patient's safety or interfere with the evaluation of the safety of PCI-24781

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Choy, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopez G, Liu J, Ren W, Wei W, Wang S, Lahat G, Zhu QS, Bornmann WG, McConkey DJ, Pollock RE, Lev DC. Combining PCI-24781, a novel histone deacetylase inhibitor, with chemotherapy for the treatment of soft tissue sarcoma. Clin Cancer Res. 2009 May 15;15(10):3472-83. doi: 10.1158/1078-0432.CCR-08-2714. Epub 2009 May 5. PMID 19417021
- [Background] Buggy JJ, Cao ZA, Bass KE, Verner E, Balasubramanian S, Liu L, Schultz BE, Young PR, Dalrymple SA. CRA-024781: a novel synthetic inhibitor of histone deacetylase enzymes with antitumor activity in vitro and in vivo. Mol Cancer Ther. 2006 May;5(5):1309-17. doi: 10.1158/1535-7163.MCT-05-0442. PMID 16731764
- [Background] Adimoolam S, Sirisawad M, Chen J, Thiemann P, Ford JM, Buggy JJ. HDAC inhibitor PCI-24781 decreases RAD51 expression and inhibits homologous recombination. Proc Natl Acad Sci U S A. 2007 Dec 4;104(49):19482-7. doi: 10.1073/pnas.0707828104. Epub 2007 Nov 27. PMID 18042714
- [Background] Yang C, Choy E, Hornicek FJ, Wood KB, Schwab JH, Liu X, Mankin H, Duan Z. Histone deacetylase inhibitor PCI-24781 enhances chemotherapy-induced apoptosis in multidrug-resistant sarcoma cell lines. Anticancer Res. 2011 Apr;31(4):1115-23. PMID 21508354
- [Background] Yang C, Choy E, Hornicek FJ, Wood KB, Schwab JH, Liu X, Mankin H, Duan Z. Histone deacetylase inhibitor (HDACI) PCI-24781 potentiates cytotoxic effects of doxorubicin in bone sarcoma cells. Cancer Chemother Pharmacol. 2011 Feb;67(2):439-46. doi: 10.1007/s00280-010-1344-7. Epub 2010 May 12. PMID 20461381
- [Background] Lopez G, Torres K, Liu J, Hernandez B, Young E, Belousov R, Bolshakov S, Lazar AJ, Slopis JM, McCutcheon IE, McConkey D, Lev D. Autophagic survival in resistance to histone deacetylase inhibitors: novel strategies to treat malignant peripheral nerve sheath tumors. Cancer Res. 2011 Jan 1;71(1):185-96. doi: 10.1158/0008-5472.CAN-10-2799. Epub 2010 Nov 16. PMID 21084276
- [Background] Choy E, Flamand Y, Balasubramanian S, Butrynski JE, Harmon DC, George S, Cote GM, Wagner AJ, Morgan JA, Sirisawad M, Mani C, Hornicek FJ, Duan Z, Demetri GD. Phase 1 study of oral abexinostat, a histone deacetylase inhibitor, in combination with doxorubicin in patients with metastatic sarcoma. Cancer. 2015 Apr 15;121(8):1223-30. doi: 10.1002/cncr.29175. Epub 2014 Dec 23. PMID 25536954

RESULTS

PARTICIPANT FLOW:
Groups:
- PCI-24781 + Doxorubicin Without Mandatory GCSF: PCI-24781 + Doxorubicin without mandatory GCSF
  PCI-24781: Capsules taken orally for 5 consecutive days starting on Day 1 of each 3 week cycle
  Doxorubicin: Administered intravenously on Day 4 of each 3 week cycle
- PCI-24781 + Doxorubicin With Mandatory GCSF: PCI-24781 + Doxorubicin with mandatory GCSF
  PCI-24781: Capsules taken orally for 5 consecutive days starting on Day 1 of each 3 week cycle
  Doxorubicin: Administered intravenously on Day 4 of each 3 week cycle
Period: Overall Study
Arm/Group | PCI-24781 + Doxorubicin Without Mandatory GCSF | PCI-24781 + Doxorubicin With Mandatory GCSF
Started | 6 | 14
Completed | 6 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PCI-24781 + Doxorubicin Without Mandatory GCSF: Study participants were enrolled into two arms. Arm A administered abexinostat and doxorubicin with optional GCSF support. Arm B administered abexinostat and doxorubicin with required GCSF support to all participants. The study uses the standard 3 + 3 phase I dose escalation design. Three cohorts of 3-6 participants were enrolled in each arm and separate inter-cohort dose escalations were performed in up to three cohorts of 3-6 participants enrolled sequentially until the maximum tolerated dose (MTD) of the combination abexinostat with doxorubicin, without (Arm A) mandatory G-CSF support was established.
- PCI-24781 + Doxorubicin With Mandatory GCSF: Study participants were enrolled into two arms. Arm A administered abexinostat and doxorubicin with optional GCSF support. Arm B administered abexinostat and doxorubicin with required GCSF support to all participants. The study uses the standard 3 + 3 phase I dose escalation design. Three cohorts of 3-6 participants were enrolled in each arm and separate inter-cohort dose escalations were performed in up to three cohorts of 3-6 participants enrolled sequentially until the maximum tolerated dose (MTD) of the combination abexinostat with doxorubicin, with (Arm B) mandatory G-CSF support was established.
- Total: Total of all reporting groups
Arm/Group | PCI-24781 + Doxorubicin Without Mandatory GCSF | PCI-24781 + Doxorubicin With Mandatory GCSF | Total
Number analyzed (Participants) | 6 | 14 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (14) | 56 (14) | 54 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 8
  Male | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Time Frame: up to 30 days after starting study drugs
Population: The two groups differ in that GCSF was offered if clinically indicated in arm 1 while it was administered to all participants in arm 2.
Measure: Number; unit: mg/m2
Arm/Group | PCI-24781 + Doxorubicin Without Mandatory GCSF | PCI-24781 With Mandatory GCSF
Number analyzed (Participants) | 6 | 14
mg/m2 | 15 | 45

2. Secondary Outcome: Dose Limiting Toxicities
Description: number of patients who experienced dose limiting toxicities
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Optional GCSF | Mandatory GCSF
Number analyzed (Participants) | 6 | 14
participants | 2 | 2

3. Secondary Outcome: Number of Partial Responses (PR)
Description: number of patients who demonstrated partial response to therapy as determined by RECIST v1.0 for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Optional GCSF | Mandatory GCSF
Number analyzed (Participants) | 6 | 14
participants | 0 | 3

4. Secondary Outcome: Rate of Progression-free Survival at 6 Months in Participants Who Received PCI-24781/Doxorubicin Combination Administration.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Optional GCSF | Mandatory GCSF
Number analyzed (Participants) | 6 | 14
participants | 1 | 6

ADVERSE EVENTS:
Groups:
- PCI-24781+Dox Without Mandated GCSF: Patients in this arm were not mandated treatment with GCSF
- PCI-24781+Dox With Mandated GCSF: Patients in this are were mandated treatment with GCSF
Arm/Group | PCI-24781+Dox Without Mandated GCSF | PCI-24781+Dox With Mandated GCSF
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/14
Other Adverse Events (participants affected / at risk) | 1/6 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCI-24781+Dox Without Mandated GCSF (N=6) | PCI-24781+Dox With Mandated GCSF (N=14)
grade 3 or 4 neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
infection (Infections and infestations) | 1 (1) | 0 (0)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCI-24781+Dox Without Mandated GCSF (N=6) | PCI-24781+Dox With Mandated GCSF (N=14)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No